CLINICAL TRIAL: NCT02287571
Title: The Effects of Preoperative Skin Traction and Position Splint on Pain, Comfort and Satisfaction in Patients With Hip Fracture
Brief Title: Skin Traction Versus Position Splint in Patients With Hip Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, BETÜL TOSUN, RN, MsN, PhD, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B.10.4.İSM.4.06.68.49/
Record Dates: First submitted 2014-11-03; First posted 2014-11-10 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Hip Fractures; Complication of Traction Procedure; Pain; Splints
Keywords: comfort; satisfaction
MeSH Terms: conditions — Hip Fractures; Pain; Personal Satisfaction | interventions — Compression Bandages

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Skin traction (Active Comparator): Prior to hip fracture surgery, affected limb was wrapped with a special elastic bandage and pulled from the sole of the foot with a weight of 5-10% of total body weight of the patient (min 2.3 kg, max 4.5 kg).
  Interventions: Device: elastic bandage
- Position splint (Experimental): Prior to hip fracture surgery, position splint was applied to the affected limb in order to keep the extremity in the proper positon without any weight lifting.
  Interventions: Device: Derotation splint

INTERVENTIONS:
Device: Derotation splint — This group is the actual intervention group.
  Arms: Position splint
Device: elastic bandage — This group is the routine treatment (control) valid in the clinical practice.
  Arms: Skin traction

SUMMARY:
The aim of this prospective, randomized controlled trial is to compare the effects of preoperative skin traction and position splint on pain, comfort, complications, difficulty level of nursing interventions, satisfaction from treatment and nursing care in patients with hip fracture. The sample is comprised of 34 patients with hip fracture in each group, totally 68 patients. Skin traction and position splint were applied after block randomization. Data regarding pain, comfort, satisfaction from care, immobilization comfort, complications, time of operation and hospitalization time were collected after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Being inpatient who were planned the surgery due to the hip fracture (caput femur fracture, collum femur fracture, femur intertrochanteric fracture and subtrochanteric fracture) diagnosis in the Orthopedics and Traumatology Clinic
* Being 50 years old or more
* Patients who speak and literate in Turkish
* Patients who gave informed consent to participate in the study

Exclusion Criteria:

* Any condition that emerges an obstacle for verbal and written interaction during data collection phase
* Unable to perform written or verbal communication in Turkish
* Withdrawal from the study due to medical reasons or death, at his/her will prior to preoperative data collection
* Urgent non-elective surgery
* Physician decision that do accept the method of immobilization assigned to the patient as appropriate

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2013-03; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Pain | up to 7 days
  Pain was assessed by VAS score prior to intervention, 15, 30, 60 and 120 minutes after intervention and daily from the next morning of intervention till the surgery.
Comfort | up to 7 days
  Comfort was assessed by VAS score prior to intervention, 15, 30, 60 and 120 minutes after intervention and by Immobilization Comfort Questionnaire daily from the next morning of intervention till the surgery.
Satisfaction from the treatment | Up to 7 days
  Satisfaction from the treatment was assessed by VAS score from the next day after intervention till the surgery.

SECONDARY OUTCOMES:
Complications | Up to 7 days
  Complications (pressure ulcer, deep vein thrombosis, allergic skin reaction, pulmonary and urinary tract infection and constipation due to immobilization) were evaluated daily after intervention till the surgery.
Surgery duration | participants were followed for the duration of surgical procedure, an average of 2 hours
  Time that the surgical procedure has taken was assessed.
Hospitalization duration | participants were followed for the duration of hospital stay, an average of 2 weeks
  Time spent in the hospital till discharge was assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Betul Tosun, RN, PhD, Principal Investigator — Saglik Bilimleri Universitesi Gulhane Tip Fakultesi; Ozlem Aslan, Assoc.Prof., Study Chair — Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Locations (1):
- Gulhane Military Medical Academy, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Resch S, Bjarnetoft B, Thorngren KG. Preoperative skin traction or pillow nursing in hip fractures: a prospective, randomized study in 123 patients. Disabil Rehabil. 2005 Sep 30-Oct 15;27(18-19):1191-5. doi: 10.1080/09638280500055800. PMID 16278188
- [Background] Saygi B, Ozkan K, Eceviz E, Tetik C, Sen C. Skin traction and placebo effect in the preoperative pain control of patients with collum and intertrochanteric femur fractures. Bull NYU Hosp Jt Dis. 2010;68(1):15-7. PMID 20345356
- [Background] Endo J, Yamaguchi S, Saito M, Itabashi T, Kita K, Koizumi W, Kawaguchi Y, Asaka T, Saegusa O. Efficacy of preoperative skin traction for hip fractures: a single-institution prospective randomized controlled trial of skin traction versus no traction. J Orthop Sci. 2013 Mar;18(2):250-5. doi: 10.1007/s00776-012-0338-1. Epub 2012 Nov 28. PMID 23187429
- [Background] Rosen JE, Chen FS, Hiebert R, Koval KJ. Efficacy of preoperative skin traction in hip fracture patients: a prospective, randomized study. J Orthop Trauma. 2001 Feb;15(2):81-5. doi: 10.1097/00005131-200102000-00001. PMID 11232658
- [Background] Koval KJ, Cooley MR. Clinical pathway after hip fracture. Disabil Rehabil. 2005 Sep 30-Oct 15;27(18-19):1053-60. doi: 10.1080/09638280500056618. PMID 16278174
- [Background] Hili S, Dawe EJ, Lindisfarne EA, Stott PM. Perioperative management of elderly patients suffering a hip fracture. Br J Hosp Med (Lond). 2014 Feb;75(2):78-82. doi: 10.12968/hmed.2014.75.2.78. PMID 24521802
- [Background] Yip DK, Chan CF, Chiu PK, Wong JW, Kong JK. Why are we still using pre-operative skin traction for hip fractures? Int Orthop. 2002;26(6):361-4. doi: 10.1007/s00264-002-0387-8. Epub 2002 Jul 13. PMID 12466869
- [Background] Anderson GH, Harper WM, Connolly CD, Badham J, Goodrich N, Gregg PJ. Preoperative skin traction for fractures of the proximal femur. A randomised prospective trial. J Bone Joint Surg Br. 1993 Sep;75(5):794-6. doi: 10.1302/0301-620X.75B5.8376442.
- [Background] Handoll HH, Queally JM, Parker MJ. Pre-operative traction for hip fractures in adults. Cochrane Database Syst Rev. 2011 Dec 7;(12):CD000168. doi: 10.1002/14651858.CD000168.pub3. PMID 22161361
- [Background] Levi N. Is preoperative tibial traction responsible for peroneal nerve palsy in patients with a fractured hip? Acta Orthop Belg. 1998 Sep;64(3):273-6. PMID 9828472
- [Background] Finsen V, Borset M, Buvik GE, Hauke I. Preoperative traction in patients with hip fractures. Injury. 1992;23(4):242-4. doi: 10.1016/s0020-1383(05)80007-5. PMID 1618564
- See also: immobilization comfort questionnaire that was used to evaluate the late period comfort of hip fracture patients is based on the comfort theory which was developed by Kathy Kolcaba. — http://www.thecomfortline.com/